CLINICAL TRIAL: NCT03588416
Title: Management of Malignant Colorectal Polyps (T1) After Endoscopic Polypectomy: Follow-up vs Surgery and Analysis of Pathological Risk Factors for Lymph Nodes Metastasis. A Retrospective and Prospective Multicentric Observational Study.
Brief Title: Multicentric Study About Pathological Risk Factors for Lymph Node Metastasis in Malignant Colorectal Polyps
Acronym: POST-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dario Parini (Other)
Responsible Party: Sponsor-Investigator, Dario Parini, Principal Investigator, Azienda Ospedaliera di Perugia
Organization: Azienda Ospedaliera di Perugia (Other)
Other Study IDs: 1359CESC
Record Dates: First submitted 2018-05-28; First posted 2018-07-17 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Colorectal Cancer; Lymph Node Metastasis; Colorectal Polyp
Keywords: pT1; Polypectomy; Lymph node metastasis; Colorectal neoplasm
MeSH Terms: conditions — Colorectal Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Colorectal cancer screening showed an increased incidence of malignant colorectal polyps pT1 after endoscopic excision. Their management is not yet standardized, for the presence of histological features increasing early lymph node involvement. The literature has proposed several histopathological criteria, for which the risk of lymph node metastasis can vary (6-20%), but final data are not yet available.

Aim 1.To collect data about patients undergoing an endoscopic polypectomy with histologic finding of pT1, retrospectively and prospectively, dividing both databases into two groups, endoscopic group (EG) and surgical group (SG) Aim 2. To analyze retrospectively which pathological criteria can increase the risk of lymph node metastasis and to elaborate a prognostic score for lymph node metastatic risk Aim 3. To verify prospectively the prognostic score capacity on predicting lymph node metastasis Aim 4. To calculate the disease free survival, overall survival, local recurrence rate and distal recurrence rate and verify if there is a difference between EG and SG

According to literature, the most important histopathological criteria to establish the high risk of lymph node metastasis are:

1. Lateral margin of healthy tissue (high risk: <1mm and piecemeal polypectomy)
2. Depth of submucosa invasion (high risk: >1000 μM or sm2-sm3 for sessile polyps; Haggitt level 4 for pedunculated polyps)
3. Vascular invasion (high risk: presence)
4. Lymphatic invasion (high risk: presence)
5. Tumor budding (high risk: presence)
6. Tumor differentiation (high risk: grade G3-G4 or mucinous)

A database will be used by all participating centres for collecting clinical and pathological data. All the analyses will be centralized by the PI. Uni-multivariate analyses will be conducted at the end of data collection for retrospective arm and at 2 years of follow-up for prospective arm.

Impact: This study aimed to investigate pathological risk factors for lymph node metastasis in pT1 colorectal polyps after endoscopic polypectomy; their accurate identification could lead to improve their management, avoiding useless complementary surgery. Results could change clinical practice and reduce health-related costs.

DETAILED DESCRIPTION:
The management of malignant colorectal tumors pT1 after polypectomy is not yet standardized, for the presence of histological features increasing early lymph node involvement. Three recent meta-analysis have identified some pathological criteria influencing the risk of lymph node metastasis in early colorectal cancer, but there is not agreement in the conclusions between these articles. Because this uncertainty, the decision making criteria for this patients can be different in every Institute. Furthermore, the majority of the literature refers to surgical patients, with lack in demonstrating, at long-term, the absence of lymph nodes metastasis in patients not operated after endoscopic polypectomy.

Retrospective study:

From a retrospective period of 6 years, with at list 2 years of follow-up, all patients who underwent endoscopic polypectomy for malignant colorectal polyp pT1, will be enrolled for the study.

The patients will be divided into two groups: patients who did only the endoscopic treatment (EG), and patients who underwent complementary surgery (SG).

The most important histopathological criteria to list in the database, when available (to establish the high risk of lymph node metastasis) are as follows:

1. Lateral margin of healthy tissue (high risk: <1mm and piecemeal polypectomy)
2. Depth of submucosa invasion (high risk: >1000 μM or sm2-sm3 for sessile polyps and Haggitt level 4 for pedunculated polyps)
3. Vascular invasion (high risk: presence); method of determination (Hematoxylin & Eosin or immunohistochemical marker)
4. Lymphatic invasion (high risk: presence); method of determination (Hematoxylin & Eosin or immunohistochemical marker)
5. Tumor budding (high risk: presence)
6. Tumor differentiation (high risk: grade G3-G4 or mucinous)

Other data to be reported are as follows:

1. Demographic and clinical data for all patients
2. Decisional context (multidisciplinary group decision; single specialist decision; patient decision) and decision making criteria for complementary surgery for all patients
3. Type of surgical resection for SG, access (laparotomy, laparoscopy or transanal), site of lesion (right, transverse, left, sigmoid colon or rectum)
4. Histopathological criteria, other than the 6 high risk criteria above
5. Histopathological finding after surgical resection for SG
6. Postoperative data (hospital stay, morbidity with Clavien-Dindo's classification) for SG
7. Type and length of follow-up for all patients (EG and SG) (endoscopic surveillance, thoracic and abdominal CT scan, positron emission computed tomography (PET-CT), carcinoembryonic antigen (CEA) determination, clinical examination)

Prospective study:

According to the histological characteristics, the patients will be considered with low risk (without any histological criteria), or with high risk (with at least one of six criteria).

The histopathological criteria to consider the malignant polyps at high risk of lymph node metastasis are as follows:

1. Lateral margin of healthy tissue <1mm and piecemeal polypectomy
2. Depth of submucosa invasion >1000 μM or sm2-sm3 for sessile polyps and Haggitt level 4 for pedunculated polyps
3. Presence of vascular invasion, determined with the immunohistochemical marker CD34 or, in alternative, with Hematoxylin & Eosin
4. Presence of lymphatic invasion, determined with the immunohistochemical marker D2-40 or, in alternative, with Hematoxylin & Eosin
5. Presence of tumor budding (low and high grade)
6. Tumor differentiation grade G3-G4 or mucinous

Patients who will present at least one of these six criteria, will be considered at high risk for lymph node metastasis.

Every Institute will take an independent decision about therapeutic strategy: only endoscopic treatment (EG), or complementary surgery (SG).

To participate to the prospective study, is mandatory to obtain these 6 pathological characteristics.

It is strongly recommended a multidisciplinary discussion for all patients, in presence of at least one surgeon, one endoscopist, one pathologist and one oncologist, as well as one radiotherapist for rectal lesions.

The surgical resection for the colon can be performed with laparotomic, laparoscopic or robotic approach, based on single Institute surgical experience. For the rectum, the surgical approach (laparotomic, laparoscopic, robotic, transanal resection) will be decided by the surgical team in accordance with the multidisciplinary group, based on single Institute experience and patient clinical features.

All patients (EG and SG) have to perform within one month from diagnosis or, in any way, before the surgery for SG, a thoracic and abdominal CT scan with contrast (for staging) and CEA determination.

The histopathological finding to be reported after surgical resection for SG are as follows: number of lymph nodes, number of metastatic lymph nodes, margin distance from the site of polypectomy, local residual tumor.

Follow-up program:

* EG: colonoscopy at 6 and 12 months for colic lesions, recto-sigmoidoscopy at 6, 18 and 24 months and colonoscopy at 12 months for rectal lesions
* SG: colonoscopy at 12 months for colic lesions, recto-sigmoidoscopy at 6, 18 and 24 months and colonoscopy at 12 months for rectal lesions
* Thoracic and abdominal CT scan with contrast at 12 and 24 months
* Clinical examination and CEA determination at 6, 12, 18 and 24 months

Statistic analysis:

Retrospective study: considering a 10% prevalence of pN+ patients with pT1 colorectal tumor, including the above 6 histopathological criteria as predictors in logistic regression model, the investigators estimate to retrospectively collect data from 600 patients.

The continuous numerical data will be expressed as average and standard deviation or as median and interquartile range, if appropriate. A descriptive analysis for collected variables will be done and the pN+ prevalence will be calculated. A logistic recession model will be estimated, for evaluating the 6 histopathological criteria effect on presence of lymph node metastasis. Furthermore, the disease-free survival will be calculated with Kaplan-Meier method. A p-value < 0.05 will be considered significant. Statistic analysis will be done with Software 3.3.2 (R Foundation for Statistical Computing, Vienna, Austria).

Prospective study: the investigators want to evaluate a sensibility of 0.80 for overall histopathological criterion (i.e., patients with at least one of six criteria are considered at high risk, patients without the six criteria are at low risk), in order that the maximum estimation error does not exceed 0.10, with a 95% confidence interval. Considering a 10% prevalence of pN+ patients with pT1 colorectal tumor, including the above 6 histopathological criteria as predictors in logistic regression model, the investigators estimate to prospectively collect data from 615 patients.

The continuous numerical data will be expressed as average and standard deviation or as median and interquartile range, if appropriate. A descriptive analysis for collected variables will be done and the pN+ prevalence will be calculated. The diagnostic capacity of the overall histopathological criterion will be evaluated calculating sensibility, specificity, positive predictive value, negative predictive value and accuracy. A similar evaluation will be done for every single histopathological criterion with explorative purpose, if appropriate. A p-value < 0.05 will be considered significant. Statistic analysis will be done with Software 3.3.2 (R Foundation for Statistical Computing, Vienna, Austria).

Statement:

With the retrospective observational study, the investigators can quickly have an extended overview about the current management of endoscopic pT1, to verify if there is, in fact, decisional heterogeneity, and to analyze the pathological criteria influence in lymph nodes metastasis. The limit of retrospective study, in the other side, is data heterogeneity, but this topic is recent, and it is normal not to have uniformity between different Institutes. This problem could be solved with the prospective study, where pathological criteria are included in the protocol itself. The strong points in this prospective project are: 1) uniformity in pathological analysis, 2) without any mandatory indication for complementary surgery, in order to maintain the observational nature of the study; 3) the multidisciplinary discussion for every patient, an aspect more and more required by hospital administrations, and 4) the uniformity in follow-up, that is a feature not yet clear in the literature for endoscopic pT1. Furthermore, this prospective study can be the base to create a national register, to set up future studies on this topic, as analysis of tumor molecular characteristics.

The elaboration of this protocol followed the STROBE statement Guidelines and Explanation.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent an endoscopic colorectal polypectomy for malignant polyp pT1

Exclusion Criteria:

* Age < 18 years
* Gastrointestinal cancer previously diagnosticated or synchronous

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent an endoscopic colorectal polypectomy with pathologic diagnosis of malignant polyp pT1
Sampling Method: Probability Sample
Enrollment: 615 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-02-29 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of patients with lymph nodes metastasis in pT1 colorectal cancer | Enrollment
  The six pathological criteria will be tested as independent predictors of lymph node metastasis
Disease free survival in EG and SG and in patients with and without high risk factors | 24 months

SECONDARY OUTCOMES:
Developing a clinical prognostic score for lymph node metastasis | Enrollment
  The clinical prognostic score will be calculated from pathological criteria and clinical risk factors (i.e. sex, age, tumor localization, size)
Validating the clinical prognostic score as predictor of lymph node metastasis | Enrollment
Overall survival | 24 months
Local and distal recurrence rate in EG and SG and in high risk patients and low risk patients | 24 months
Sensitivity and specificity of diagnostic tests in detecting pathologic lymph nodes | Enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Santa Maria della Misericordia - ULSS 5 Polesana, Rovigo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mou S, Soetikno R, Shimoda T, Rouse R, Kaltenbach T. Pathologic predictive factors for lymph node metastasis in submucosal invasive (T1) colorectal cancer: a systematic review and meta-analysis. Surg Endosc. 2013 Aug;27(8):2692-703. doi: 10.1007/s00464-013-2835-5. Epub 2013 Feb 8. PMID 23392988
- [Background] Beaton C, Twine CP, Williams GL, Radcliffe AG. Systematic review and meta-analysis of histopathological factors influencing the risk of lymph node metastasis in early colorectal cancer. Colorectal Dis. 2013 Jul;15(7):788-97. doi: 10.1111/codi.12129. PMID 23331927
- [Background] Wada H, Shiozawa M, Katayama K, Okamoto N, Miyagi Y, Rino Y, Masuda M, Akaike M. Systematic review and meta-analysis of histopathological predictive factors for lymph node metastasis in T1 colorectal cancer. J Gastroenterol. 2015 Jul;50(7):727-34. doi: 10.1007/s00535-015-1057-0. Epub 2015 Mar 1. PMID 25725617
- [Background] Haggitt RC, Glotzbach RE, Soffer EE, Wruble LD. Prognostic factors in colorectal carcinomas arising in adenomas: implications for lesions removed by endoscopic polypectomy. Gastroenterology. 1985 Aug;89(2):328-36. doi: 10.1016/0016-5085(85)90333-6. PMID 4007423
- [Background] Kikuchi R, Takano M, Takagi K, Fujimoto N, Nozaki R, Fujiyoshi T, Uchida Y. Management of early invasive colorectal cancer. Risk of recurrence and clinical guidelines. Dis Colon Rectum. 1995 Dec;38(12):1286-95. doi: 10.1007/BF02049154. PMID 7497841
- [Background] Ueno H, Murphy J, Jass JR, Mochizuki H, Talbot IC. Tumour 'budding' as an index to estimate the potential of aggressiveness in rectal cancer. Histopathology. 2002 Feb;40(2):127-32. doi: 10.1046/j.1365-2559.2002.01324.x. PMID 11952856
- [Background] van de Velde CJ, Boelens PG, Borras JM, Coebergh JW, Cervantes A, Blomqvist L, Beets-Tan RG, van den Broek CB, Brown G, Van Cutsem E, Espin E, Haustermans K, Glimelius B, Iversen LH, van Krieken JH, Marijnen CA, Henning G, Gore-Booth J, Meldolesi E, Mroczkowski P, Nagtegaal I, Naredi P, Ortiz H, Pahlman L, Quirke P, Rodel C, Roth A, Rutten H, Schmoll HJ, Smith JJ, Tanis PJ, Taylor C, Wibe A, Wiggers T, Gambacorta MA, Aristei C, Valentini V. EURECCA colorectal: multidisciplinary management: European consensus conference colon & rectum. Eur J Cancer. 2014 Jan;50(1):1.e1-1.e34. doi: 10.1016/j.ejca.2013.06.048. Epub 2013 Oct 31. PMID 24183379
- [Background] Bartel MJ, Brahmbhatt BS, Wallace MB. Management of colorectal T1 carcinoma treated by endoscopic resection from the Western perspective. Dig Endosc. 2016 Apr;28(3):330-41. doi: 10.1111/den.12598. Epub 2016 Feb 16. PMID 26718885
- [Background] Steele SR, Chang GJ, Hendren S, Weiser M, Irani J, Buie WD, Rafferty JF; Clinical Practice Guidelines Committee of the American Society of Colon and Rectal Surgeons. Practice Guideline for the Surveillance of Patients After Curative Treatment of Colon and Rectal Cancer. Dis Colon Rectum. 2015 Aug;58(8):713-25. doi: 10.1097/DCR.0000000000000410. PMID 26163950
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Epidemiology. 2007 Nov;18(6):800-4. doi: 10.1097/EDE.0b013e3181577654. PMID 18049194
- [Background] Vandenbroucke JP, von Elm E, Altman DG, Gotzsche PC, Mulrow CD, Pocock SJ, Poole C, Schlesselman JJ, Egger M; STROBE Initiative. Strengthening the Reporting of Observational Studies in Epidemiology (STROBE): explanation and elaboration. Epidemiology. 2007 Nov;18(6):805-35. doi: 10.1097/EDE.0b013e3181577511. PMID 18049195